CLINICAL TRIAL: NCT02606383
Title: Non-inferiority, Phase III Clinical Trial Comparing Dapaconazole Cream 2% (Biolab Sanus Farmacêutica Ltda.) Versus Ketoconazole Cream 2% (Nizoral® Janssen-Cilag) in Patients With Tinea Pedis
Brief Title: Non-inferiority Phase III Trial Comparing Dapaconazole Cream 2% With Ketoconazole Cream 2% in Patients With Tinea Pedis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDN 007/15
Record Dates: First submitted 2015-11-12; First posted 2015-11-17 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — 1-(2-(2,4-dichlorophenyl)-2-(4-(trifluoromethyl)benzyloxy)ethyl)-1H-imidazole; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapaconazole (Experimental): Dapaconazole 2% Cream Topical
  Interventions: Drug: Dapaconazole
- Ketoconazole (Active Comparator): Ketoconazole 2% Cream Topical
  Interventions: Drug: Ketoconazole

INTERVENTIONS:
Drug: Dapaconazole
  Other Names: BL123
  Arms: Dapaconazole
Drug: Ketoconazole
  Arms: Ketoconazole

SUMMARY:
This is a non-inferiority, Phase III, open-label, randomized, parallel trial to evaluate the new intervention Dapaconazole cream 2% versus Ketoconazole cream 2% in patients with Tinea pedis. Sample size is 140 participants (70 per treatment group), male or female, aged between 16 and 60 years-old.

Primary objective is to evaluate non-inferiority of Dapaconazole cream 2% compared to Ketoconazole cream 2% in Tinea pedis treatment. Secondary objective is to evaluate safety and tolerability of Dapaconazole cream 2% after multiple administrations.

Participants will receive either new intervention or active control during 14 consecutive days, which will be followed by 2 follow-up visits.

Primary efficacy endpoint is clinical and mycological lesion cure, and secondary efficacy endpoint is time (days) until clinical diagnosis of lesion cure. Additionally, safety will be assessed by adverse events occurrence and laboratory exams evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female study participants, aged between 16 and 60 years-old. Patients aged between 16 and 18 years-old will provide additional Assent Form before enrollment in the trial;
* Presence of a skin lesion characteristic of Tinea pedis, with diagnosis confirmed by direct mycological exam;
* Absence of previous antifungic treatment for the lesion under study;
* Absence of other significant diseases which, at the physician's discretion, could have an impact on subject's participation in the trial, according to protocol requirements, and study evaluations: medical history, blood pressure and heart rate measurements, physical examination and screening laboratory tests;
* Ability to understand the nature and objectives of the trial, including risks and adverse events; willingness to cooperate with the researcher and proceed according to all study requirements, which shall be confirmed by Informed Consent Form signature.

Exclusion Criteria:

* Known hypersensitivity to ketoconazole or chemically related compounds; history of serious adverse reactions;
* Screening laboratory tests results showing clinically relevant deviations that, at the researcher discretion, prevent the subject to participate in the trial due to possible risks;
* Drugs addiction, including alcohol;
* Use of any previous treatment to the lesion under study that, according to principal investigator best judgement, might interfere in study objectives;
* Treatment, within 3 months before the trial, with any drugs known to have a well-established toxic potential to major organs;
* Participation in any other experimental research or administration of any experimental drug within 6 months before this trial;
* Pregnancy, labor or miscarriage with 12 weeks before study treatment;
* Any conditions, according to investigator's best judgement, that prevents the subject to participate in the trial.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Clinical cure of the lesion | 14 days
  Assessment of presence or absence of the lesion by clinical examination
Mycological cure of the lesion | 14 days
  Laboratory test for presence or absence of Tinea pedis

SECONDARY OUTCOMES:
Time (days) until clinical diagnosis of lesion cure | 14 days

OTHER OUTCOMES:
Safety and tolerability | 45 days
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, PhD, Principal Investigator — Galeno Desenvolvimento de Pesquisas Ltda.
Locations (1):
- Clínica Gobbato de Dermatologia, Rio Claro, São Paulo, Brazil